CLINICAL TRIAL: NCT01704105
Title: WASH Benefits Kenya: A Cluster Randomized Controlled Trial of the Benefits of Sanitation, Water Quality, Handwashing, and Nutrition Interventions on Child Health and Development
Brief Title: WASH Benefits Kenya
Acronym: WASHB-Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovations for Poverty Action (Other)
Collaborators: Kenya Medical Research Institute (Other); University of California, Berkeley (Other); University of California, Davis (Other); Tufts University (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Clair Null, Research Affiliate, Innovations for Poverty Action
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IPA-2012-KE; 2011-09-3654 (Other: UC Berkeley)
Record Dates: First submitted 2012-10-05; First posted 2012-10-11 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Malnutrition; Diarrhea; Child Development
Keywords: Chlorine water treatment; Point-of-use water treatment; Household water treatment with safe storage; Handwashing with soap; Hand hygiene; Latrines; Water; Sanitation; Handwashing; Breast Feeding; Complementary Feeding; Micronutrients; Malnutrition; Nutrition Disorders; Diarrhea; Child Development; Child potties; Point-of-use fortification; Lipid-based nutrient supplement; Exclusive breastfeeding; Environmental enteropathy; Tropical enteropathy; Gut function; Intestinal parasitic infection; Soil transmitted helminths; Intestinal protozoans; Antibody response
MeSH Terms: conditions — Malnutrition; Diarrhea; Breast Feeding; Nutrition Disorders; Sprue, Tropical; Intestinal Diseases, Parasitic | interventions — Water Quality; Sanitation; Hand Disinfection; Nutritional Status

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Analysts and lab technicians were masked to intervention status. Outcome collectors were not informed of intervention status, but could have inferred status from observing intervention hardware during household visits.
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Water Quality (Active Comparator): 100 clusters, approximately 1,000 newborns
  Interventions: Behavioral: Water Quality
- Sanitation (Active Comparator): 100 clusters, approximately 1,000 newborns
  Interventions: Behavioral: Sanitation
- Handwashing (Active Comparator): 100 clusters, approximately 1,000 newborns
  Interventions: Behavioral: Handwashing
- Combined Water, Sanitation, and Handwashing (Active Comparator): 100 clusters, approximately 1,000 newborns
  Interventions: Behavioral: Water Quality; Behavioral: Sanitation; Behavioral: Handwashing
- Nutrition (Active Comparator): 100 clusters, approximately 1,000 newborns
  Interventions: Dietary Supplement: Nutrition
- Nutrition + Combined Water, Sanitation, and Handwashing (Active Comparator): 100 clusters, approximately 1,000 newborns
  Interventions: Behavioral: Water Quality; Behavioral: Sanitation; Behavioral: Handwashing; Dietary Supplement: Nutrition
- Active control arm (No Intervention): 200 clusters, approximately 2,000 newborns. Village-level promoter will visit household and will strictly engage in recording the child's MUAC, which will also be conducted in all active comparator arms as well.
- Passive control arm (No Intervention): 100 clusters, approximately 1,000 newborns. No intervention.

INTERVENTIONS:
Behavioral: Water Quality — Hardware: Chlorine dispensers provided for free at communal water sources. Promotion: Local promoters will visit study compounds at least monthly during the first year and bi-monthly thereafter to deliver behavior change messages that focus on the treatment of drinking water for all children living in the household.
  Arms: Combined Water, Sanitation, and Handwashing; Nutrition + Combined Water, Sanitation, and Handwashing; Water Quality
Behavioral: Sanitation — Hardware: Free child potties, sani-scoop hoes to remove feces from household environments, and new or upgraded pit latrine for each study compound. Upgrades may include structural improvements, plastic slabs, and superstructure improvements.
  Promotion: Local promoters will visit study compounds at least monthly during the first year and bi-monthly thereafter to deliver behavior change messages that focus on the use of latrines for defecation and the removal of human and animal feces from the compound.
  Arms: Combined Water, Sanitation, and Handwashing; Nutrition + Combined Water, Sanitation, and Handwashing; Sanitation
Behavioral: Handwashing — Hardware: Handwashing "dual tippy tap" stations, including jugs for clean and for soapy water. Handwashing stations will be stocked with soap for the duration of the trial.
  Promotion: Local promoters will visit study compounds at least monthly during the first year and bi-monthly thereafter to deliver behavior change messages that focus on handwashing with soap at critical times around food preparation, defecation, and contact with feces.
  Arms: Combined Water, Sanitation, and Handwashing; Handwashing; Nutrition + Combined Water, Sanitation, and Handwashing
Dietary Supplement: Nutrition — Supplement: Lipid-based Nutrient Supplement (LNS) twice daily from ages 6 to 24 months.
  Promotion: Local promoters will visit study compounds at least monthly during the first year and bi-monthly thereafter to deliver behavior change messages modeled on those recommended in the Guiding Principles for Complementary Feeding of the Breastfed Child and the recent UNICEF Program Guide for Infant and Young Child Feeding Practices. General messages will include (1) practice exclusive breastfeeding from birth to 6 months of age and introduce complementary foods at 6 months of age while continuing to breastfeed; (2) continue breast feeding as you did before receiving LNS; (3) provide your child micronutrient-rich foods such as meat, fish, eggs, and vitamin A rich fruits and vegetables; and (4) feed your child at least 2-3 times per day when 6-8 months old and 3-4 times per day when 9-24 months old.
  Arms: Nutrition; Nutrition + Combined Water, Sanitation, and Handwashing

SUMMARY:
The purpose of this study is to measure the independent and combined effects of interventions that improve sanitation, water quality, handwashing, and nutrition on child health and development in the first years of life.

DETAILED DESCRIPTION:
Children in resource-poor settings are at risk of multiple episodes of diarrhea, enteric infections, and environmental enteropathy, an inflammatory disorder of the intestines that compromises nutrient absorption (1). In cross-sectional analyses, repeated episodes of diarrhea and chronic environmental enteropathy in early childhood are associated with reduced growth and cognitive function, and impaired school performance which can reduce income later in life (2-8). Although more evidence is needed to establish causal links, repeated episodes of childhood diarrhea and enteric infection may exact a long-run toll, perpetuating a cycle of poverty and ill health.

Infection and inadequate diet are proximate risk factors for undernutrition and early life growth faltering; the two processes likely act reciprocally in a vicious cycle that perpetuates physiologic and metabolic deficits and increases the risk of mortality. Children who exhibit growth faltering are more likely to have deficits in cognitive development and long-term human capital, and are more likely to have children who also suffer from growth deficits - perpetuating the cycle into the next generation.

There are two probable interdependent pathways that link enteric infections to child growth and development. The first pathway includes repeated infections that lead to acute illness or parasitic infection in the first years of life, which increase the risk of stunting and subsequent cognitive deficits in childhood and later in life. The second pathway is through subclinical environmental enteropathy.

There is limited evidence to demonstrate whether or not water quality, sanitation, and handwashing (WASH) interventions can improve measures of environmental enteropathy, child growth and development, and whether nutritional interventions could be enhanced if provided concurrently with WASH interventions. To help fill this evidence gap, the WASH Benefits study will deliver randomized interventions designed to reduce infection and improve nutrition, and will measure intervention effects on child illness, growth and development. WASH Benefits includes two, comparable but standalone trials in Bangladesh and Kenya that are registered under separate protocols.

In Kenya, the study will include approximately 800 clusters, and each cluster will enroll approximately 10 household compounds with pregnant women in their second or third trimester. The study will randomize 100 clusters to each of 6 active intervention arms (water quality, sanitation, handwashing, combined WSH, nutrition, nutrition+WSH), 200 clusters to a double size active control arm, and 100 clusters to a single-sized passive control arm (measurement pending future funding). Children born into the cohort will be followed for 2 years after the intervention, with measurements at 12 and 24 months after intervention delivery. (anticipated age range: 20 - 27 months old at the final measurement). At the 12- and 24-month follow-up visits, the study will collect child anthropometric measurements and caregiver-reported diarrhea. In the final visit the study will administer a test to measure child development outcomes. The study will collect urine, blood, and stool specimens from a subsample of 1,500 children distributed across four arms of the study (Active Control, Combined WSH, Nutrition, Nutrition+WSH) to measure biomarkers of gut function and intestinal parasitic infections at the 12- and 24-month follow-up visits. In addition, the study will collect specimens (blood, stool) from children 18 - 27 months old at baseline who are living in the same compound as target children to test for intestinal parasitic infections.

ELIGIBILITY:
Study Population Description:

The subject population will be young children and their mothers/guardians living in several contiguous districts of Western Province, in the rural areas outside the towns of Bungoma and Kakamega. Communities must meet the following criteria:

* Located in a rural area (defined as villages with <25% residents living in rental houses, <2 gas/petrol stations and <10 shops)
* Not enrolled in ongoing WASH or nutrition programs
* No chlorine dispensers at water sources installed by programs separate from the present study
* Majority (>80%) of households do not have access to piped water into the home
* At least six eligible pregnant women in the cluster at baseline.

From enrolled communities, household compounds will be enrolled if they meet the following criteria.

Inclusion Criteria:

1. One or more women who self-identify as pregnant at the time of the baseline survey
2. The woman plans to stay in the community for the next 12 months.

Exclusion Criteria:

(1) The study excludes households who do not own their home to help mitigate attrition during follow-up.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8246 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Length-for-Age Z-scores | Measured 24 months after intervention
  Child's recumbent length, standardized to Z-scores using the WHO 2006 growth standards, measured 24 months after intervention. Measurement techniques follow the FANTA 2003 protocol.
Diarrhea Prevalence | Measured 12 and 24 months after intervention
  Diarrhea is defined as 3+ loose or watery stools in 24 hours or 1+ stools with blood in 24 hours. Diarrhea will be measured in interviews using caregiver-reported symptoms with 2-day and 7-day recall, measured 12 and 24 months after intervention.

SECONDARY OUTCOMES:
Length-for-Age Z-scores | Measured 12 months after intervention
  Child's recumbent length, standardized to Z-scores using the WHO 2006 growth standards, measured 12 months after intervention. Measurement techniques follow the FANTA 2003 protocol
Stunting Prevalence | Measured 24 months after intervention
  Child's recumbent length, standardized to Z-scores using the WHO 2006 growth standards, measured 24 months after intervention. Measurement techniques follow the FANTA 2003 protocol. Children with length-for-age Z-scores < - 2 will be classified as stunted.
Enteropathy Biomarkers | Measured 12- and 24 months after intervention
  The lactulose / mannitol dual sugar permeability test will be administered to children. The ratio of the recovery of the two sugars in the urine will be used to calculate the L:M ratio, and we will compare groups using logged values of the ratio. We will measure myeloperoxidase, alpha 1-antitrypsin, and neopterin levels in the stool. We will additionally measure Total IgG antibody titers in the blood, and we will compare groups using logged values of the antibody levels.
ASQ Child Development Scores | Measured 24 months after intervention
  Interviewers will administer a locally adapted version of the Ages and Stages Questionnaire (ASQ) to children after 24 months of intervention. The ASQ includes item sets of caregiver-reported milestones that measure child development in three separate domains (gross motor, communication, personal/social skills).

OTHER OUTCOMES:
Infection with ascaris, trichuris, hookworm, and giardia | Measured 24 months after interventions began
  Infection with soil transmitted helminths (ascaris, trichuris, hookworm) will be enumerated in stool collected from all index children and one older child per study compound. Giardia will also be measured in stool samples collected form these children. Prevalence and eggs per gram of feces will be recorded.
Hemoglobin concentration and anemia | Measured 24 months after interventions began
  Hemoglobin concentrations will be measured using venous blood samples with a Hemocue 301 analyzer.
Micronutrient status, including iron, vitamin A, folate, and B12 | Measured 24 months after interventions began
  Iron status will be assessed using the biomarkers of ferritin, soluble transferrin receptor (sTfR), and hepcidin. Vitamin A status will be assessed using retinol binding protein. Folate and B12 status will be measured using plasma folate and B12.

CONTACTS AND LOCATIONS:
Overall Officials: Clair Null, PhD, Principal Investigator — Innovations for Poverty Action and Mathematica Policy Research; Christine Stewart, PhD, Principal Investigator — University of California, Davis; Amy Pickering, PhD, Principal Investigator — Tufts University
Locations (1):
- Innovations for Poverty Action, Kenya, Kisumu, P.O Box 2663, Kenya

REFERENCES:
- [Background] Haghighi P, Wolf PL. Tropical sprue and subclinical enteropathy: a vision for the nineties. Crit Rev Clin Lab Sci. 1997;34(4):313-41. doi: 10.3109/10408369708998096. PMID 9288443
- [Background] Borghi J, Guinness L, Ouedraogo J, Curtis V. Is hygiene promotion cost-effective? A case study in Burkina Faso. Trop Med Int Health. 2002 Nov;7(11):960-9. doi: 10.1046/j.1365-3156.2002.00954.x. PMID 12390603
- [Background] Alderman H, Hoddinott J, Kinsey B. Long term consequences of early childhood malnutrition. Oxford Economic Papers-New Series 2006;58:450-474.
- [Background] Checkley W, Buckley G, Gilman RH, Assis AM, Guerrant RL, Morris SS, Molbak K, Valentiner-Branth P, Lanata CF, Black RE; Childhood Malnutrition and Infection Network. Multi-country analysis of the effects of diarrhoea on childhood stunting. Int J Epidemiol. 2008 Aug;37(4):816-30. doi: 10.1093/ije/dyn099. Epub 2008 Jun 20. PMID 18567626
- [Background] Lorntz B, Soares AM, Moore SR, Pinkerton R, Gansneder B, Bovbjerg VE, Guyatt H, Lima AM, Guerrant RL. Early childhood diarrhea predicts impaired school performance. Pediatr Infect Dis J. 2006 Jun;25(6):513-20. doi: 10.1097/01.inf.0000219524.64448.90. PMID 16732149
- [Background] Niehaus MD, Moore SR, Patrick PD, Derr LL, Lorntz B, Lima AA, Guerrant RL. Early childhood diarrhea is associated with diminished cognitive function 4 to 7 years later in children in a northeast Brazilian shantytown. Am J Trop Med Hyg. 2002 May;66(5):590-3. doi: 10.4269/ajtmh.2002.66.590. PMID 12201596
- [Background] Petri WA Jr, Miller M, Binder HJ, Levine MM, Dillingham R, Guerrant RL. Enteric infections, diarrhea, and their impact on function and development. J Clin Invest. 2008 Apr;118(4):1277-90. doi: 10.1172/JCI34005. PMID 18382740
- [Background] Boissiere M, Knight JB, Sabot RH. Earnings, schooling, ability, and cognitive skills. American Economic Review 1985;75:1016-1030.
- [Derived] Stewart CP, Arnold CD, Williams AM, Arnold BF, Pickering AJ, Dentz H, Kiprotich M, Lin A, Null C, Colford JM Jr, Dewey KG. Social Desirability Bias in a Randomized Controlled Trial That Included Breastfeeding Promotion in Western Kenya. Curr Dev Nutr. 2024 Sep 23;9(Suppl 1):103779. doi: 10.1016/j.cdnut.2024.103779. eCollection 2025 Feb. PMID 40454163
- [Derived] Pickering AJ, Njenga SM, Steinbaum L, Swarthout J, Lin A, Arnold BF, Stewart CP, Dentz HN, Mureithi M, Chieng B, Wolfe M, Mahoney R, Kihara J, Byrd K, Rao G, Meerkerk T, Cheruiyot P, Papaiakovou M, Pilotte N, Williams SA, Colford JM Jr, Null C. Effects of single and integrated water, sanitation, handwashing, and nutrition interventions on child soil-transmitted helminth and Giardia infections: A cluster-randomized controlled trial in rural Kenya. PLoS Med. 2019 Jun 26;16(6):e1002841. doi: 10.1371/journal.pmed.1002841. eCollection 2019 Jun. PMID 31242190
- [Derived] Stewart CP, Dewey KG, Lin A, Pickering AJ, Byrd KA, Jannat K, Ali S, Rao G, Dentz HN, Kiprotich M, Arnold CD, Arnold BF, Allen LH, Shahab-Ferdows S, Ercumen A, Grembi JA, Naser AM, Rahman M, Unicomb L, Colford JM Jr, Luby SP, Null C. Effects of lipid-based nutrient supplements and infant and young child feeding counseling with or without improved water, sanitation, and hygiene (WASH) on anemia and micronutrient status: results from 2 cluster-randomized trials in Kenya and Bangladesh. Am J Clin Nutr. 2019 Jan 1;109(1):148-164. doi: 10.1093/ajcn/nqy239. PMID 30624600
- [Derived] Byrd KA, Williams TN, Lin A, Pickering AJ, Arnold BF, Arnold CD, Kiprotich M, Dentz HN, Njenga SM, Rao G, Colford JM Jr, Null C, Stewart CP. Sickle Cell and alpha+-Thalassemia Traits Influence the Association between Ferritin and Hepcidin in Rural Kenyan Children Aged 14-26 Months. J Nutr. 2018 Dec 1;148(12):1903-1910. doi: 10.1093/jn/nxy229. PMID 30517728
- [Derived] Stewart CP, Kariger P, Fernald L, Pickering AJ, Arnold CD, Arnold BF, Hubbard AE, Dentz HN, Lin A, Meerkerk TJ, Milner E, Swarthout J, Colford JM Jr, Null C. Effects of water quality, sanitation, handwashing, and nutritional interventions on child development in rural Kenya (WASH Benefits Kenya): a cluster-randomised controlled trial. Lancet Child Adolesc Health. 2018 Apr;2(4):269-280. doi: 10.1016/S2352-4642(18)30025-7. PMID 29616236
- [Derived] Null C, Stewart CP, Pickering AJ, Dentz HN, Arnold BF, Arnold CD, Benjamin-Chung J, Clasen T, Dewey KG, Fernald LCH, Hubbard AE, Kariger P, Lin A, Luby SP, Mertens A, Njenga SM, Nyambane G, Ram PK, Colford JM Jr. Effects of water quality, sanitation, handwashing, and nutritional interventions on diarrhoea and child growth in rural Kenya: a cluster-randomised controlled trial. Lancet Glob Health. 2018 Mar;6(3):e316-e329. doi: 10.1016/S2214-109X(18)30005-6. Epub 2018 Jan 29. PMID 29396219
- [Derived] Williams AM, Stewart CP, Shahab-Ferdows S, Hampel D, Kiprotich M, Achando B, Lin A, Null CA, Allen LH, Chantry CJ. Infant Serum and Maternal Milk Vitamin B-12 Are Positively Correlated in Kenyan Infant-Mother Dyads at 1-6 Months Postpartum, Irrespective of Infant Feeding Practice. J Nutr. 2018 Jan 1;148(1):86-93. doi: 10.1093/jn/nxx009. PMID 29378045
- [Derived] Williams AM, Chantry CJ, Young SL, Achando BS, Allen LH, Arnold BF, Colford JM Jr, Dentz HN, Hampel D, Kiprotich MC, Lin A, Null CA, Nyambane GM, Shahab-Ferdows S, Stewart CP. Vitamin B-12 Concentrations in Breast Milk Are Low and Are Not Associated with Reported Household Hunger, Recent Animal-Source Food, or Vitamin B-12 Intake in Women in Rural Kenya. J Nutr. 2016 May;146(5):1125-31. doi: 10.3945/jn.115.228189. Epub 2016 Apr 13. PMID 27075905
- [Derived] Arnold BF, Null C, Luby SP, Unicomb L, Stewart CP, Dewey KG, Ahmed T, Ashraf S, Christensen G, Clasen T, Dentz HN, Fernald LC, Haque R, Hubbard AE, Kariger P, Leontsini E, Lin A, Njenga SM, Pickering AJ, Ram PK, Tofail F, Winch PJ, Colford JM Jr. Cluster-randomised controlled trials of individual and combined water, sanitation, hygiene and nutritional interventions in rural Bangladesh and Kenya: the WASH Benefits study design and rationale. BMJ Open. 2013 Aug 30;3(8):e003476. doi: 10.1136/bmjopen-2013-003476. PMID 23996605
- See also: Click here for more information about this study — http://www.washbenefits.net
- See also: Related protocol — http://www.clinicaltrials.gov/ct2/show/NCT01590095